CLINICAL TRIAL: NCT02783885
Title: Clinical Utilization of Newly Approved Oncology Medications in Middle Eastern Population
Brief Title: Clinical Utilization of Newly Approved Oncology Medications
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Guard Health Affairs (Other Government)
Responsible Party: Sponsor
Other Study IDs: RC15/097/R
Record Dates: First submitted 2016-05-12; First posted 2016-05-26 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: immunotherapy

SUMMARY:
The efficacy and safety of different medications vary from one individual to another and from one ethnic group to another. Therefore, strong interest in the study of pharmacogenomic and pharmacoepidemiology has evolved recently.

There are multiple examples of oncology drugs being more effective in certain ethnic population compared to other. For example, irinotecan combined with cisplatin was very effective drug in the management of small cell lung cancer in the Japanese patients while an identical study done in the US revealed no major benefit to this combination in American population

DETAILED DESCRIPTION:
Another example is having more benefit drawn from tyrosine kinase inhibitors (Erlotinib or Gefitinib) in Asian patients.

Immunotherapy is a new class of cancer treatment that works to harness the innate powers of the immune system to fight cancer. Because of the immune system's unique properties, these therapies may hold greater potential than current treatment approaches to fight cancer more powerfully, to offer longer-term protection against the disease, to come with fewer side effects, and to benefit more patients with more cancer types

Immunotherapy includes treatments that work in different ways. Some boost the body's immune system in a very general way. Others help train the immune system to attack cancer cells specifically. Immunotherapy has become an important part of treating some types of cancer. Newer types of immune treatments are now being studied, and they'll impact how we treat cancer in the future.

Recently, multiple immunotherapy treatment been approved with a couple of EGFR resistant medications.

Many new oncology drugs are being used in Middle Eastern countries including Saudi Arabia for different indications without being studied in the Middle Eastern population. These medications' efficacy and safety profiles may differ from those patients studied for drug development and approval due to difference in population's characteristics.

The goal of this study is to observe, summarize and report the patterns of the use of these drugs and describe their efficacy and safety profile in the early phases of their use.

The investigators aim is to build on the existing experience and knowledge by utilization of classic methodology and approaches on a larger scale and more effective way to paint picture of the performance of a certain therapy in the real life world. The use of prospective design will help evaluate the efficacy and safety of therapies already used in practice, generate new hypothesis, and/or determine the outcome of certain diseases.

ELIGIBILITY:
Inclusion Criteria:

* All patients with cancer or hematological malignancies receiving new oncology medications (defined as a medication in the first five years of their introduction to the ME market
* Patient accepts to participate in study and signing consent form

Exclusion Criteria:

* None

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oncology centers managing patients with solid tumors or hematological malignancies in the national Guard and the investigators can open it in other Middle Eastern countries if the investigators need more sample size as Tawam Hospital (UAE), Alhamad Hospital (Qatar), AUB (Lebanon) and Algeria
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-05; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Descriptive measures of the pattern of use of the new medications in our population | 3 years

SECONDARY OUTCOMES:
Measuring the efficacy in terms of response | 3 years
Measuring the efficacy in terms of progression-free survival (PFS) | 3 years
Measuring the efficacy in terms of overall survival (OS) | 3 years

CONTACTS AND LOCATIONS:
Locations (2):
- Saudi Arabia (2):
  - King Abdul Aziz Medical City for National Guard Health Affairs, Riyadh
  - King Abdul Aziz Medical City for National Guard, Riyadh

IPD SHARING:
Plan to Share IPD: No